CLINICAL TRIAL: NCT04566588
Title: Early Apical Release vs Classic Holmium Laser Enucleation of the Prostate: Randomized Controlled Trial Comparing Post-Operative Incontinence Rates and Surgical Outcomes
Acronym: HoLEP EAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Don Neff, MD, FACS, Associate Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 145490
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early apical release holmium enucleation of the prostate (Experimental): Early apical release holmium enucleation of the prostate (EAR HoLEP), as a surgical treatment for benign prostatic hyperplasia
  Interventions: Procedure: EAR HoLEP
- Classic holmium enucleation of the prostate (Active Comparator): Classic holmium enucleation of the prostate (HoLEP), as a surgical treatment for benign prostatic hyperplasia
  Interventions: Procedure: Classic HoLEP

INTERVENTIONS:
Procedure: EAR HoLEP — early apical release holmium enucleation of the prostate (EAR HoLEP), as a surgical treatment for benign prostatic hyperplasia
  Arms: Early apical release holmium enucleation of the prostate
Procedure: Classic HoLEP — classic holmium enucleation of the prostate as a surgical treatment for benign prostatic hyperplasia
  Arms: Classic holmium enucleation of the prostate

SUMMARY:
To determine if early apical release holmium enucleation of the prostate (EAR HoLEP), as a surgical treatment for benign prostatic hyperplasia, reduces post-operative urinary incontinence compared to classic HoLEP.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older
* Patients must present to clinic with a diagnosis of benign prostatic hyperplasia
* Patients must be scheduled to undergo a holmium laser enucleation of the prostate

Exclusion Criteria:

* Patients with previous surgical management of BPH
* Patients with prostate biopsy revealing high risk prostate cancer
* Patients with a concomitant neurogenic bladder diagnosis (SCI, Parkinson, MS, cerebral palsy)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Post-operative Urinary Incontinence | Twelve Months Post-operative
  to determine if patients who undergo early apical release HoLEP have reduced rates of post-operative urinary incontinence compared to classic HoLEP as measured by patient report of leakage

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Health System, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No